CLINICAL TRIAL: NCT02649569
Title: Continuous Activity Monitoring During Fractionated Radiotherapy: A Pilot Study
Brief Title: Continuous Activity Monitoring During Fractionated Radiotherapy in Patients With Head and Neck, Lung, or Gastrointestinal Cancer
Status: Completed | Type: Observational
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nitin Ohri, Principal Investigator, Albert Einstein College of Medicine
Other Study IDs: 2015-4873; NCI-2015-02292 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 007067; 2015-4873 (Other: Albert Einstein College of Medicine); P30CA013330 (NIH)
Record Dates: First submitted 2016-01-06; First posted 2016-01-07 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Digestive System Carcinoma; Head and Neck Carcinoma; Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Monitoring, Physiologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational (continuous activity monitoring, questionnaires): Patients wear an activity monitor throughout and up 4 weeks after completion of radiation therapy. Patients who are willing may continue to wear the monitor through routine follow up appointments. Patients also complete questionnaires at evaluations, which take place prior to radiotherapy initiation, weekly during radiotherapy, and then 2 and 4 weeks after the completion of radiotherapy.
  Interventions: Device: Monitoring Device; Other: Quality-of-Life Assessment

INTERVENTIONS:
Device: Monitoring Device — Wear activity monitor
  Other Names: Monitor
Other: Quality-of-Life Assessment — Complete the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30
  Other Names: Quality of Life Assessment

SUMMARY:
This pilot research trial studies continuous activity monitoring during fractionated radiotherapy in patients with head and neck, lung, or gastrointestinal cancer. This study explores the use of fitness trackers to study the activity levels of patients before, during, and after radiation therapy and the use of weekly assessments to measure the patients' quality of life during radiation therapy. This may allow doctors to see if there is any relationship between activity levels, quality of life, treatment interruptions, hospitalizations, and clinical outcomes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate the feasibility of continuous, accelerometer-based evaluation of patient activity levels before, during, and after treatment with fractionated external beam radiotherapy.

SECONDARY OBJECTIVES:

I. To demonstrate the feasibility of performing weekly quality of life assessments during fractionated external beam radiotherapy.

II. To explore how accelerometer-based metrics change throughout patients' treatment courses and if these changes are associated with quality of life assessments, treatment interruptions, hospitalizations, and clinical outcomes.

OUTLINE:

Patients wear an activity monitor throughout and up 4 weeks after completion of radiation therapy. Patients who are willing may continue to wear the monitor through routine follow up appointments. Patients also complete questionnaires at evaluations, which take place prior to radiotherapy initiation, weekly during radiotherapy, and then 2 and 4 weeks after the completion of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Able to ambulate independently (without the assistance of a cane or walker)
* Diagnosis of invasive malignancy of the head and neck region, lung, or gastrointestinal tract
* Planned treatment with fractionated (>= 15 treatments) external beam radiotherapy with concurrent chemotherapy with curative intent
* Women of childbearing potential must:

  * Have a negative serum or urine pregnancy test within 72 hours prior to the start of study therapy
  * Agree to utilize an adequate method of contraception throughout treatment and for at least 4 weeks after study therapy is completed
  * Be advised of the importance of avoiding pregnancy during trial participation and the potential risks of an unintentional pregnancy
* All patients must sign study specific informed consent prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Planned treatment with fractionated (>= 15 treatments) external beam radiotherapy with concurrent chemotherapy with curative intent
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2015-06; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Number of patients who complete most (>= 80%) of the protocol-specified assessments | Up to 4 weeks post-chemoradiation therapy
  This pilot study will yield preliminary data on the feasibility of activity monitoring during radiotherapy as well as possible associations between activity level and various clinical and treatment-related variables. Data from the study will be summarized using standard descriptive statistics; means and standard deviations will be used for normally-distributed continuous variables, and frequencies and percentages will be used for categorical variables. Exploratory analyses for associations between activity levels and clinical and treatment-related variables will be performed using chi-square o
Number of patients who successfully use the activity monitor (i.e. wearing the activity monitor throughout the treatment course) | Up to 4 weeks post-chemoradiation therapy
  This pilot study will yield preliminary data on the feasibility of activity monitoring during radiotherapy as well as possible associations between activity level and various clinical and treatment-related variables. Data from the study will be summarized using standard descriptive statistics; means and standard deviations will be used for normally-distributed continuous variables, and frequencies and percentages will be used for categorical variables. Exploratory analyses for associations between activity levels and clinical and treatment-related variables will be performed using chi-square o

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Ohri, Principal Investigator — Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - Albert Einstein College of Medicine, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York